CLINICAL TRIAL: NCT01271660
Title: A Randomized, Double-blinded, Placebo-controlled Study Evaluating the Efficacy and Safety of 6-week Treatment of Pregabalin Against Frequent Muscle Cramp in Patients With Liver Cirrhosis
Brief Title: A Study Evaluating the Efficacy and Safety of Pregabalin Against Frequent Muscle Cramp in Patients With Liver Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Boramae Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Won Kim, MD, PhD, Assistant Professor, Seoul National University Boramae Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-2010-132; IG-KOR-014-2010 (Other: Pfizer reference number)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Muscle Cramp; Liver Cirrhosis
Keywords: muscle cramp; liver cirrhosis; pregabalin
MeSH Terms: conditions — Muscle Cramp; Liver Cirrhosis | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Active Comparator): 30 randomly allocated patients after a 4-week run-in period, who will take part in a 6-week treatment period with pregabalin.
  Treatment period : 75 mg twice daily during the first 1 week as titration + 150mg twice daily for 4 weeks as standard dose period + 75mg twice a day for a week as tapering period.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): 30 randomly allocated patients after a 4-week run-in period, who will take part in a 6-week treatment period with placebo.
  Treatment period : 75 mg twice daily during the first 1 week as titration + 150mg twice daily for 4 weeks as standard dose period + 75mg twice a day for a week as tapering period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — drug form : capsule, 75/150mg. Pregabalin will be provided to treatment arm subjects for 6-week Treatment period.
  Treatment period : 75 mg twice daily during the first 1 week as titration + 150mg twice daily for 4 weeks as maintenance + 75mg twice a day as tapering
  Other Names: Brand name of drug : Lyrica
  Arms: Pregabalin
Drug: Placebo — drug form : capsule, 75/150mg. Pregabalin will be provided to treatment arm subjects for 6-week Treatment period.
  Treatment period : 75 mg twice daily during the first 1 week as titration + 150mg twice daily for 4 weeks as maintenance + 75mg twice a day as tapering
  Arms: Placebo

SUMMARY:
Muscle cramp is defined as a paroxysmal, involuntary, and painful contraction of skeletal muscle. Cirrhotic patients can encounter with muscle cramp frequently, which might be associated with poor quality of life. Gabapentin can be prescribed for muscle cramp. However, patients with liver cirrhosis have limited access to gabapentin which is metabolized primarily in liver.

Pregabalin with a similar mechanism of action to gabapentin undergoes negligible metabolism owing to its improved pharmacokinetic properties. Thus, pregabalin might be a promising therapeutic option for patients with liver cirrhosis who are suffering from muscle cramp and susceptible to drug-induced hepatotoxicity.

Therefore, the investigators hypothesize that pregabalin could effectively reduce painful symptoms derived from muscle cramp. In the current study, the investigators are going to evaluate the efficacy and safety of pregabalin by comparing outcomes between two groups (treatment group vs. placebo group).

DETAILED DESCRIPTION:
The investigators are planning to recruit patients with liver cirrhosis and muscle cramp, and collect the baseline clinical and laboratory data during the 4-week run-in period for each subject. After a run-in period, there will be the second step of patient selection to achieve a more homogenous study population. Then, patients will be randomly allocated into the treatment (pregabalin) and placebo (dummy) arms, by a web-based randomization program. After a treatment period (75 mg twice daily during the first 1 week as titration, 150 mg twice daily for 4 weeks as standard dose), the investigators will gather further study information of a standard dose period (150mg twice daily for 4 weeks) from the target population and the study subjects will enter the 1-week tapering period (75mg twice a day) to discontinuation. The primary outcome will be the difference in the frequency of muscle cramps between the run-in and treatment phases. The investigators also intend to assess the response rate, defined as the proportion (%) of patients showing ≥50% reduction in the number of muscle cramps, mean change in the average pain intensity, mean change in the score of the Short Form 36 (SF-36, QualityMetric) health survey questionnaire, mean change in the frequency of muscle cramps during sleep, and mean change in the average cramp threshold frequency by the neurophysiologic study (nerve excitability test) and analyze the reasons for drop-out cases.

ELIGIBILITY:
Inclusion Criteria: (should follow all conditions described below)

* Etiology : Liver cirrhosis patients of any etiology, whether viral or non-viral
* Occurrence of muscle cramp equal to or more than 2 times a week over the last month

Exclusion Criteria:

* Preexisting disease : Occlusive vascular disease, thyroid disease, peripheral neuropathy
* Drugs within 2 months : Digitalis, cimetidine, clofibrate, lithium, opiate, nifedipine, beta-agonist, beta-blocker, penicillamine, gabapentin, pregabalin, tricyclic anti-depressant, carbamazepine, phenytoin, quinidine, antispastic drugs, verapamil, vitamin E, branched chain amino acid, excessive alcohol consumption (male >40 g/day, female >20 g/day)
* Underlying disease : Renal impairment (Ccr < 60 mL/min), neuromuscular disease (stroke, cerebral palsy, multiple sclerosis, Parkinson disease, progressive muscular dystrophy, epilepsy), suicidal attack, drug allergy, pregnancy, heart failure
* Liver status : Serious complications resulting from decompensated cirrhosis except ascites, such as portosystemic encephalopathy, acute variceal bleeding within the past 3 months from study entry
* central nervous system (CNS) or peripheral nervous system (PNS) or muscular disease, stroke, cerebral palsy, multiple sclerosis, Parkinson disease, progressive muscular dystrophy, epilepsy
* The previous episode of suicidal attack
* Drug hypersensitivity
* Subjects receiving antiepileptic drugs
* Patients manipulating machines or driving cars
* Pregnant women
* Subjects with congestive heart failure requiring medications
* Galactose-Lactose metabolic abnormality
* Refractory ascites to medical treatment

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Difference in the frequency of muscle cramps between run-in and treatment phases (/week) | after 4 weeks of standard dose treatment period
  The frequency is defined as muscle cramps per week.

SECONDARY OUTCOMES:
Response rates , Mean change in the average cramp pain intensity , peripheral nerve excitability , the quality of life, quality of sleep , safety | after 4 weeks of standard dose treatment period or over a 6-week treatment period
  Response rates : the proportion (%) of patients showing ≥50% reduction in the number of muscle cramps.
  Mean change in the average cramp pain intensity : a sum of the pain rating scale divided by a total number of muscle cramps.
  Peripheral nerve excitability as measured by nerve stimulation test.
  The quality of life as measured by mean change in the score of the SF-36.
  Quality of sleep as measured by mean change in the number of muscle cramps during sleep.
  Safety as measured by dose-reduction or discontinuation rates, treatment-emergent adverse events, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Won Kim, Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahn S, Hong YH, Lee DH, Joo SK, Jung YJ, Sohn SY, Choi K, Kim W. Efficacy and Safety of Pregabalin for Muscle Cramps in Liver Cirrhosis: A Double-Blind Randomized Controlled Trial. J Korean Med Sci. 2022 Feb 21;37(7):e56. doi: 10.3346/jkms.2022.37.e56. PMID 35191232